CLINICAL TRIAL: NCT03792932
Title: A Multicenter Prospective RCT Study of Laparoscopic Versus Open Distal Pancreatectomy in Patients With Pancreatic Cancer at the Body and Tail
Brief Title: Laparoscopic vs Open Pancreatectomy for Body and Tail Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Chair of Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPAC-2
Record Dates: First submitted 2018-12-27; First posted 2019-01-04 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Pancreatic Cancer; Surgery; Laparoscopy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laparoscopic distal pancreatectomy (Active Comparator)
  Interventions: Procedure: Laparoscopic distal pancreatectomy
- Open distal pancreatectomy (Active Comparator)
  Interventions: Procedure: Open distal pancreatectomy

INTERVENTIONS:
Procedure: Laparoscopic distal pancreatectomy — Laparoscopic distal pancreatectomy includes distal pancreatectomy, splenectomy, and regional lymph nodes resection for pancreatic cancer at the body and tail. Regional lymph nodes includes group 8, 10, 11, 18, 7, 9, 14, 15, according to the 2003 edition of lymph nodes group system defined by Japan Pancreas Society (JPS).
  Arms: Laparoscopic distal pancreatectomy
Procedure: Open distal pancreatectomy — Open distal pancreatectomy includes distal pancreatectomy, splenectomy, and regional lymph nodes resection for pancreatic cancer at the body and tail. Regional lymph nodes includes group 8, 10, 11, 18, 7, 9, 14, 15, according to the 2003 edition of lymph nodes group system defined by Japan Pancreas Society (JPS).
  Arms: Open distal pancreatectomy

SUMMARY:
Open distal pancreatectomy (ODP) has been commonly employed for the treatment of a variety of cancers in body and tail of pancreas. Although many general surgical procedures have been increasingly performed laparoscopically or with laparoscopic assistance, until the current decade, laparoscopic pancreatic surgery had not been performed for its complicated anatomy. But laparoscopic distal pancreatectomy (LDP) has been widely accepted as a standard treatment for body and tail pancreatic cancer because there is no anastomosis in it, and LDP has gradually become the first choice for these cancers in clinical work. Although there are several studies about the comparison between LDP and ODP, most are retrospective and there is no agreement in surgical margin, lymph node numbers and prognosis to identify the oncological differences between the two surgical approaches. The investigators' pilot study showed that patients with body and tail pancreatic cancer underwent LDP had a better prognosis compared with the ones undergoing ODP, with no statistics differences in postoperative complications and mortality. This perspective RCT study is performed to confirm whether LDP would improve the prognosis for patients with body and tail pancreatic cancer compared with ODP.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years and ≤ 80 years, no gender limitation
2. Resectable body and tail pancreatic cancer (refer to NCCN 2018)
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
4. Tumor locates at the body and tail of the pancreas without distant metastasis
5. No celiac trunk and superior mesenteric artery invasion
6. No operation contraindication, fit for laparoscopic surgery
7. The expected survival after surgery ≥ 3 months
8. Patients who are willing and able to comply with the study procedure
9. Signed informed content obtained prior to treatment

Exclusion Criteria:

1. Locally advanced unresectable body and tail pancreatic cancer
2. Multi-organ and vascular resection needed
3. Patients undergoing total pancreatectomy
4. Benign tumor at the body and tail of the pancreas or pancreatic cancer at the head of the pancreas
5. Distant metastasis or ascites detected by imaging
6. Severe important organ function impairment (heart, liver, kidney)
7. Patients who are with other primary malignancy or haematological disorders
8. Pregnant or nursing women
9. Patients who have received chemotherapy, radiotherapy and interventional therapy before the pancreatectomy
10. Patients who have participated in other clinical trials for pancreatic cancer treatment within 3 months

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2019-02-02 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival | 2 years
  RFS

SECONDARY OUTCOMES:
Overall Survival | 2 years
  OS
R0 resection rate | 2 years
  R0 resection rate
Detected lymph node number | 2 years
  Detected lymph node number

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui
  - Department of Hepatobiliary and Pancreatic Surgery, The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Department of Hepatopancreatobiliary Surgery, Second Affiliated Hospital of Harbin Medical University,, Harbin, Heilongjiang
  - Department of Biliary-Pancreatic Surgery, Affiliated Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Department of Hepato-Pancreato-Biliary Surgery, The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Shanghai Pancreatic Cancer Institute; Pancreatic Cancer Institute, Fudan University. Shanghai, China, Shanghai, Shanghai Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan
  - Department of Gastroenterology and Pancreatic Surgery, Zhejiang Provincial People's Hospital, Hanzhou, Zhejiang
  - Department of Pancreatic and Biliary Surgery, The First Affiliated Hospital of Harbin Medical University, Harbin
  - Department of Biliopancreatic Surgery, Huadong Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ricci C, Casadei R, Taffurelli G, Toscano F, Pacilio CA, Bogoni S, D'Ambra M, Pagano N, Di Marco MC, Minni F. Laparoscopic versus open distal pancreatectomy for ductal adenocarcinoma: a systematic review and meta-analysis. J Gastrointest Surg. 2015 Apr;19(4):770-81. doi: 10.1007/s11605-014-2721-z. Epub 2015 Jan 6. PMID 25560180
- [Background] van Hilst J, de Rooij T, Klompmaker S, Rawashdeh M, Aleotti F, Al-Sarireh B, Alseidi A, Ateeb Z, Balzano G, Berrevoet F, Bjornsson B, Boggi U, Busch OR, Butturini G, Casadei R, Del Chiaro M, Chikhladze S, Cipriani F, van Dam R, Damoli I, van Dieren S, Dokmak S, Edwin B, van Eijck C, Fabre JM, Falconi M, Farges O, Fernandez-Cruz L, Forgione A, Frigerio I, Fuks D, Gavazzi F, Gayet B, Giardino A, Groot Koerkamp B, Hackert T, Hassenpflug M, Kabir I, Keck T, Khatkov I, Kusar M, Lombardo C, Marchegiani G, Marshall R, Menon KV, Montorsi M, Orville M, de Pastena M, Pietrabissa A, Poves I, Primrose J, Pugliese R, Ricci C, Roberts K, Rosok B, Sahakyan MA, Sanchez-Cabus S, Sandstrom P, Scovel L, Solaini L, Soonawalla Z, Souche FR, Sutcliffe RP, Tiberio GA, Tomazic A, Troisi R, Wellner U, White S, Wittel UA, Zerbi A, Bassi C, Besselink MG, Abu Hilal M; European Consortium on Minimally Invasive Pancreatic Surgery (E-MIPS). Minimally Invasive versus Open Distal Pancreatectomy for Ductal Adenocarcinoma (DIPLOMA): A Pan-European Propensity Score Matched Study. Ann Surg. 2019 Jan;269(1):10-17. doi: 10.1097/SLA.0000000000002561. PMID 29099399
- [Background] Sulpice L, Farges O, Goutte N, Bendersky N, Dokmak S, Sauvanet A, Delpero JR; ACHBT French Pancreatectomy Study Group. Laparoscopic Distal Pancreatectomy for Pancreatic Ductal Adenocarcinoma: Time for a Randomized Controlled Trial? Results of an All-inclusive National Observational Study. Ann Surg. 2015 Nov;262(5):868-73; discussion 873-4. doi: 10.1097/SLA.0000000000001479. PMID 26583678
- [Background] Shin SH, Kim SC, Song KB, Hwang DW, Lee JH, Lee D, Lee JW, Jun E, Park KM, Lee YJ. A comparative study of laparoscopic vs. open distal pancreatectomy for left-sided ductal adenocarcinoma: a propensity score-matched analysis. J Am Coll Surg. 2015 Feb;220(2):177-85. doi: 10.1016/j.jamcollsurg.2014.10.014. Epub 2014 Oct 31. PMID 25529901
- [Background] Venkat R, Edil BH, Schulick RD, Lidor AO, Makary MA, Wolfgang CL. Laparoscopic distal pancreatectomy is associated with significantly less overall morbidity compared to the open technique: a systematic review and meta-analysis. Ann Surg. 2012 Jun;255(6):1048-59. doi: 10.1097/SLA.0b013e318251ee09. PMID 22511003